CLINICAL TRIAL: NCT03780218
Title: Evaluation of Pulmonary Function and Respiratory Muscle Strength in Patients With Burn Injury.
Brief Title: Evaluation of Pulmonary Function in Burn Injury
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ozden Ozkal, Principal Investigator, Hacettepe University
Other Study IDs: GO 18/1110
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2018-12

CONDITIONS: Burns
Keywords: Burn Injury; Pulmonary function; Respiratory muscle; Peripheral muscle
MeSH Terms: conditions — Burns | interventions — Inhalation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group:Respiratory function: Patients with burn injury will be included in this study. Their respiratory functions will be evaluated. Pulmonary function test, respiratory muscle strength and peripheral muscle strength will be assessed on the discharge week.
  Interventions: Other: Respiratory function
- Control Group:Respiratory function: Healthy subjects will be included in this study.Their respiratory functions will be evaluated. Pulmonary function test, respiratory muscle strength and peripheral muscle strength will be assessed.
  Interventions: Other: Respiratory function

INTERVENTIONS:
Other: Respiratory function — Respiratory function test evaluates the participants' pulmonary function and respiratory muscle strength

SUMMARY:
This study evaluates the pulmonary function, respiratory muscle strength and peripheral muscle strength in patients with burn injury on the week that they will be discharge from the hospital. Healthy subjects will be evaluated for pulmonary function, respiratory muscle strength and peripheral muscle strength.

DETAILED DESCRIPTION:
Burn injures have adverse effect on the respiratory system.In addition to burn injury prolonged hospitalization may increase the ratio of respiratory complications. But, there are no information in the literature about pulmonary function, respiratory muscle strength and peripheral muscle strength in patients with burn injury. Especially, when the patients are discharged from the hospital, it is not known whether the patients are at the same level in terms of pulmonary functions respiratory muscle strength and peripheral muscle strength with healthy individuals. This study will assess pulmonary functions respiratory muscle strength and peripheral muscle strength in patients with burn injury compared to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Having a burn injury
* Treatment by an inpatient
* able and willing to complete the informed consent process.
* Control group consists of healthy adults with the similar demographic characteristics as experimental group

Exclusion Criteria:

* having a pulmonary system disease
* having a cardiac system disease
* to do regular sports for the last three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experimental group: Patients with burn injury Control Group: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity | 15 minutes
  is the total amount of air exhaled during the test. After three trial, the best forced vital capacity value is the outcome
Forced Expiratory Volume in 1 Second | 15 minutes
  Forced Expiratory Volume in 1 Second is the volume exhaled during the first second of a forced expiratory maneuver started from the level of total lung capacity. After three trial, the best FVC value is the outcome.
Forced Expiratory Volume in 1 Second / Forced Vital Capacity | 15 minutes
  The ratio of Forced Expiratory Volume in 1 Second / Forced Vital Capacity. This formule is calculated by measuring device. After three trial, the best value is the outcome.
Maximal Inspiratory Pressure | 15 minutes
  is a measure of the strength of inspiratory muscles, primarily the diaphragm. It is obtained by having the patient inhale as strongly as possible against a mouthpiece. After three trial, the best value is the outcome.
Maximal Expiratory Pressure | 15 minutes
  a measure of the strength of respiratory muscles, obtained by having the patient exhale as strongly as possible against a mouthpiece. After three trial, the best value is the outcome.

SECONDARY OUTCOMES:
Peak Expiratory Flow | 15 minutes
  Peak Expiratory Flow is a person's maximum speed of expiration, as measured with a peak flow meter, a small, hand-held device used to monitor a person's ability to breathe out air. After three trial, the best value is the outcome.
forced expiratory flow | 15 minutes
  Forced expiratory flow is the flow (or speed) of air coming out of the lung during the middle portion of a forced expiration.
Peripheral strength | 15 minutes
  Peripheral (Grip) strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles
Pain severity | 15 minutes
  Pain severity was assessed by visual analogue scale. This scale score range from "no pain=0 point " to "worst imaginable pain=10 points" for intensity. Maximum point means worst pain severity.
Functional Exercise Capacity | 10 minutes
  It was evaluated by six minutes walk test.The 6-min walk test is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The distance will be recorded. The higher distance is indicated better exercise capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Ozkal, Principal Investigator — Hacettepe University
Locations (1):
- Ozden Ozkal, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozkal O, Topuz S, Karahan S, Erdem MM, Konan A, Yasti AC. Clinical predictors of pulmonary functions, respiratory/peripheral muscle strength and exercise capacity at discharge in adults with burn injury. Disabil Rehabil. 2021 Oct;43(20):2875-2881. doi: 10.1080/09638288.2020.1720320. Epub 2020 Jan 30. PMID 31999499